CLINICAL TRIAL: NCT04459858
Title: GTA-The Influence of the Greater Tuberosity Angle on the Clinical Outcome One Year Postoperative in Patients With a Rotator Cuff Tear - a Comparative Study.
Brief Title: The Influence of the Greater Tuberosity Angle on the Clinical Outcome One Year Postoperative in Patients With a Rotator Cuff Tear
Acronym: GTA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01201; ch20Taha2
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Rotator Cuff Tear
Keywords: Critical Shoulder Angle (CSA); Greater Tuberosity Angle (GTA)
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rotator cuff lesion: patients treated for traumatic or degenerative rotator cuff lesion
  Interventions: Other: data analysis

INTERVENTIONS:
Other: data analysis — Data is extracted from the existing medical records and from the Rotator Cuff Repair Database (RCR_USB). The GTA (determined as the angle between a "line parallel to the humerus diaphysis passing through the humeral head center of rotation and a line connecting the upper border of the humeral head to the most superolateral edge of the greater tuberosity") is determined.

SUMMARY:
This retrospective study is to investigate the influence of the Greater Tuberosity Angle (GTA) in addition to CSA on patient outcome in patients with rotator cuff tear.

DETAILED DESCRIPTION:
A tear of the rotator cuff is one of the most common disorders of the shoulder. It is assumed that a large Critical Shoulder Angle (CSA) is associated with the occurrence of rotator cuff tears. This retrospective study is to investigate the influence of the Greater Tuberosity Angle (GTA) in addition to CSA on patient outcome in patients with rotator cuff tear.

ELIGIBILITY:
Inclusion Criteria:

* Patient after an arthroscopic rotator cuff repair
* 1 to 4 years postoperative
* Presence of pre-operative radiography of the shoulder

Exclusion Criteria:

* Massive irreparable cuff tear
* Chronically retracted tendons and atrophic rotator cuff muscles Partial arthroscopic repair
* Absence of pre-operative radiography in neutral rotation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for traumatic or degenerative rotator cuff lesion at the University Hospital Basel between January 2015 and January 2019.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Constant Score | 1 year (before surgery and 1 year after surgery)
  This scoring system consists of four variables that are used to assess the function of the shoulder. The right and left shoulders are assessed separately.
  The subjective variables are pain and activity of daily life (ADL) (sleep, work, recreation / sport) which give a total of 35 points. The objective variables are range of motion and strength which give a total of 65 Points (the higher the score the better the shoulder function).

CONTACTS AND LOCATIONS:
Overall Officials: Mohy Taha, Dr. med., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland